CLINICAL TRIAL: NCT01352247
Title: Total or Partial Knee Arthroplasty Trial
Acronym: TOPKAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0606/88; ISRCTN03013488 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2011-04-20; First posted 2011-05-11 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unicompartmental Knee Replacement (Experimental): TOPKAT will be pragmatic in terms of implant selection for the knee replacement operation. Providing the inclusion criteria are met, surgeons will be entirely free to use an implant of their choice or will use the current implants used at their institution. Implant type used on each patient will be recorded.
  A partial knee replacement or UKR involves only the diseased area of the joint being replaced. The healthy compartment of the knee is retained and artificial implants are inserted in place of the diseased area. This is done via a minimally invasive surgical procedure.
  Interventions: Procedure: Unicompartmental Knee Replacement
- Total Knee Replacement (Experimental): TOPKAT will be pragmatic in terms of implant selection for the knee replacement operation. Providing the inclusion criteria are met, surgeons will be entirely free to use an implant of their choice or will use the current implants used at their institution. Implant type used on each patient will be recorded.
  A total knee replacement involves all surfaces of the knee being replaced. The procedure involves excising both diseased and normal femoral condyles, the tibial plateau and often the patella. This is done through a large skin incision which provides easy access to the knee joint. Each component will be replaced with an artificial implant, which may be cemented in position.
  Interventions: Procedure: Total Knee Replacement

INTERVENTIONS:
Procedure: Unicompartmental Knee Replacement — A partial knee replacement or UKR involves only the diseased area of the joint being replaced. The healthy compartment of the knee is retained and artificial implants are inserted in place of the diseased area. This is done via a minimally invasive surgical procedure.
  Arms: Unicompartmental Knee Replacement
Procedure: Total Knee Replacement — A total knee replacement involves all surfaces of the knee being replaced. The procedure involves excising both diseased and normal femoral condyles, the tibial plateau and often the patella. This is done through a large skin incision which provides easy access to the knee joint. Each component will be replaced with an artificial implant, which may be cemented in position.
  Arms: Total Knee Replacement

SUMMARY:
In the majority of patients with osteoarthritis of the knee the disease originates in the medial compartment. There are two different approaches to replacing this arthritic area. Some surgeons feel that it is always best to replace both the knee compartments with a Total Knee Replacement (TKR). Others feel it is best to replace just the damaged component of the knee with a Unicompartmental Knee Replacement (UKR). There is little agreement amongst knee surgeons. Both interventions are established and well documented procedures, yet little evidence exists to support either practice. Each intervention is considered standard care. There exists little evidence, however, to prove the clinical and cost effectiveness of either management option.

The aim of the Total or Partial Knee Arthroplasty Trial (TOPKAT) will be to assess the clinical and cost effectiveness of Total Knee Replacements versus Unicompartmental Knee Replacements in patients with medial osteoarthritis. This will be examined using an appropriate patient base and long term assessments.

The trial has a combined device/expertise based allocation depending on the local situation. Surgeons who are in equipoise and have sufficient experience to perform both TKR and UKR, randomisation and allocation can be based on "device" (UKR or TKR). The same surgeon will perform the operation for both arms of the study.

For surgeons who hold a preference for one treatment over the other, an "expertise" based randomisation will then occur. UKR surgeons will work alongside TKR surgeons. Patients recruited to the study from these sites will be randomised to one of the treatment options and treated by the appropriate surgeon. In such cases the patient is internally referred to the other surgeon's operating list.

Patients will be recruited by their consultant knee surgeons in collaboration with the local research team. TOPKAT are hoping to recruit 500 patients altogether, with 250 per arm of the trial.

DETAILED DESCRIPTION:
The design of the study is a single layer multicentre superiority type randomised controlled trial of unilateral knee replacement patients. The randomised controlled trial design will help reduce and prevent potential bias influencing the evaluation.

Participants will be randomised to either UKR or TKR. The trial has a combined equipoise/expertise approach. It enables surgeons who are not in equipoise to deliver only one of the two operations while also allowing surgeons in equipoise to provide both operations. A surgeon who is in equipoise ('equipoise surgeon') and has sufficient experience to perform both TKR and UKR will deliver the allocated operation (UKR or TKR). The same surgeon will perform the operation for both arms of the study.

Not all surgeons are able to exhibit this equipoise. They may hold a preference for one treatment over the other often due to experience/expertise with one type of operation. Interestingly, a surgeon may also believe the patient may benefit from one particular operation even though they may not be able to perform it themselves.

Equipoise is difficult to investigate or establish. Self declaration has been used as the main approach but in order to sufficiently secure this state the following aspects are important:

* The equipoise considered must be patient- or individual-based equipoise rather than an overall or general category equipoise based on operation type. The surgeon must consider their position for each individual patient. Only if they believe that either operation will be suitable for an individual patient can the patient then be recruited.
* No surgeon will ever knowingly perform what they consider a substandard surgical procedure.

In order to complete the trial by seeking to maximise surgeon participation, an 'expertise'-based delivery of the intervention will also occur. For this approach there must be a surgeon with expertise in TKR and a surgeon with expertise in UKR in the same centre who will act together as a 'delivery unit'. Patients recruited to the study who are under the care of such a surgeon ('expertise surgeon') will be randomised to one of the two groups and treated by the appropriate surgeon. This 'expertise' approach allows for those UKR surgeons who work alongside TKR surgeons to team up and participate in the study. Subsequent surgery may be carried out by a surgeon different to that at the initial consultation. In such cases the patient is internally referred to the other surgeon's operating list. No restriction is made upon the number of delivery units within a centre. A surgeon can only be in one delivery unit, that is, they are either an 'equipoise surgeon' or an 'expertise surgeon'.

ELIGIBILITY:
Inclusion Criteria

* Medial compartment osteoarthritis with exposed bone on both femur and tibia
* Functionally intact Anterior Cruciate Ligament (superficial damage or splitting is acceptable)
* Full thickness and good quality lateral cartilage present
* Correctable intra-articular varus deformity (suggestive of functionally intact medical cruciate ligament)
* Medically fit showing an American Society of Anesthesiologists (ASA) of 1 or 2

Exclusion Criteria

* Require revision knee replacement surgery
* Have rheumatoid arthritis or other inflammatory disorders
* Are unlikely to be able to perform required clinical assessment tasks
* Have symptomatic foot, hip or spinal pathology
* Previous knee surgery other than diagnostic arthroscopy and medial menisectomy
* Previously had septic arthritis
* Have significant damage to the patella-Femoral Joint especially on the lateral facet.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Pain and Function | Year 5 (additional extended follow-up to 10 years)
  This will be measured by using the Oxford Knee Score, a patient reported outcome questionnaire.

SECONDARY OUTCOMES:
Range of Motion and Function | Year 5
  This will be measured using the American Knee Society Score (AKSS). A clinician assessed score examining pain, stability, range of movement and function.
Activity level | Year 5 (additional extended follow-up to 10 years)
  This will be measured using two patient reported questionnaires, the University of California, Los Angeles (UCLA) Activity Score and the High Activity Arthroplasty Score.
Economic Evaluation | Year 5 (additional extended follow-up to 10 years)
  The EuroQol (EQ-5D) a patient reported questionnaire will provide data for economic evaluation.
Patient Satisfaction | Year 5 (additional extended follow-up to 10 years)
  Patient satisfaction will be measured using the Lund Score.

CONTACTS AND LOCATIONS:
Overall Officials: David Beard, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre NHS Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beard DJ, Davies LJ, Cook JA, MacLennan G, Price A, Kent S, Hudson J, Carr A, Leal J, Campbell H, Fitzpatrick R, Arden N, Murray D, Campbell MK. Total versus partial knee replacement in patients with medial compartment knee osteoarthritis: the TOPKAT RCT. Health Technol Assess. 2020 Apr;24(20):1-98. doi: 10.3310/hta24200. PMID 32369436
- [Result] Beard DJ, Davies LJ, Cook JA, MacLennan G, Price A, Kent S, Hudson J, Carr A, Leal J, Campbell H, Fitzpatrick R, Arden N, Murray D, Campbell MK; TOPKAT Study Group. The clinical and cost-effectiveness of total versus partial knee replacement in patients with medial compartment osteoarthritis (TOPKAT): 5-year outcomes of a randomised controlled trial. Lancet. 2019 Aug 31;394(10200):746-756. doi: 10.1016/S0140-6736(19)31281-4. Epub 2019 Jul 17. PMID 31326135
- [Derived] Beard DJ, Davies LJ, Cook JA, MacLennan G, Hudson J, Price AJ, Carr AJ, Little M, Leal J, Fitzpatrick R, Murray DW, Campbell MK; TOPKAT Study Group. Assessing clinical and cost effectiveness of total versus partial knee replacement (TOPKAT): 10-year follow-up of a multicentre, randomised controlled trial. Lancet Rheumatol. 2025 Nov 18:S2665-9913(25)00250-4. doi: 10.1016/S2665-9913(25)00250-4. Online ahead of print. PMID 41270774
- [Derived] Patel R, Tilling K, Lawlor DA, Howe LD, Bogdanovich N, Matush L, Nicoli E, Kramer MS, Martin RM. Socioeconomic differences in childhood length/height trajectories in a middle-income country: a cohort study. BMC Public Health. 2014 Sep 8;14:932. doi: 10.1186/1471-2458-14-932. PMID 25200513
- [Derived] Beard D, Price A, Cook J, Fitzpatrick R, Carr A, Campbell M, Doll H, Campbell H, Arden N, Cooper C, Davies L, Murray D. Total or Partial Knee Arthroplasty Trial - TOPKAT: study protocol for a randomised controlled trial. Trials. 2013 Sep 12;14:292. doi: 10.1186/1745-6215-14-292. PMID 24028414
- See also: Trial Website — https://w3.abdn.ac.uk/hsru/topkat/
- See also: Surgical Intervention Trials Unit (SITU): Coordinating Centre — https://www.situ.ox.ac.uk/surgical-trials/total-or-partial-knee-arthoplasty-trial-topkat